CLINICAL TRIAL: NCT07365436
Title: Study for Imaging the Lower Gastrointestinal Tract Using a Colonoscopy-Compatible OCT Probe
Brief Title: Imaging the Colon Using a Colonoscope Compatible Imaging Probe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025P001541; 1R01CA280972-01A1 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Colon Polyps; Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Undergoing Colorectal Screening (Experimental): 250 adult participants undergoing colorectal screening will be enrolled at MGH.
  Interventions: Device: Feasibility of using a CC-OCT probe to image the GI tract

INTERVENTIONS:
Device: Feasibility of using a CC-OCT probe to image the GI tract — 250 participants will be enrolled in this study. All consented participants will receive the same intervention.

SUMMARY:
The goal of this study is to use a colonoscope compatible device capable of taking images of the lower gastrointestinal tract. The main question it aims to answer is:

Is the colonoscope compatible optical coherence tomography probe (CC-OCT probe) an effective device to use to take images of the gut?

During the participant's standard of care colonoscopy, the CC-OCT probe will be inserted into the colonoscope. The CC-OCT probe will then collect images of the participant's gastrointestinal tract in real time.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older
* Capable of giving informed consent
* Capable of following bowel prep instructions

Exclusion Criteria:

* 75 years of age or older
* Any contraindication to bowel prep or colonoscopy
* Current diagnosis of any bleeding disorders
* Currently using drugs that interfere with coagulation (excluding low-dose aspirin)
* Pregnancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Ability of the CC-OCT to image the lower GI tract | Images are collected during the study procedure and analyzed within one year of collection

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, M.D., PhD, Principal Investigator — Massachusetts General Hospital